CLINICAL TRIAL: NCT06229028
Title: Examining the Effects of Patient Information Forms, Exercise Forms and Video Recordings on Clinical and Functional Results in Patients With Hand and Forearm Injuries.
Brief Title: Examining the Effects of Patient Information Forms, Exercise Forms and Video Recordings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, HANDE USTA, Assistant Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-60116787-020-468698
Record Dates: First submitted 2024-01-09; First posted 2024-01-29 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Hand Injuries; Work-related Injury
Keywords: hand injuries; leaflet; functional outcome
MeSH Terms: conditions — Hand Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- verbal explanation group (Experimental): The treatment by the diagnosis will be explained under the guidance of the therapist and will be repeated at each appointment to the first group.
  Interventions: Other: hand rehabilitation with verbal explanation
- patient information and exercise forms group (Experimental): Treatment by the diagnosis will be provided with patient information and exercise forms containing visual and written information in addition to an explanation under the guidance of the therapist for the second group.
  Interventions: Other: hand rehabilitation with patient information and exercise forms
- video recording group (Experimental): Treatment by diagnosis will be provided with patient information containing visual and written information, exercise forms, and video recording, in addition to narration under the guidance of the therapist for the third group.
  Interventions: Other: hand rehabilitation with video recording

INTERVENTIONS:
Other: hand rehabilitation with verbal explanation — Patients in all groups will undergo a 12-week hand rehabilitation process that includes the use of appropriate orthoses if necessary, approaches to edema and pain, restoration of joint range of motion, strengthening, and functional return to work or activities. The application of the rehabilitation process will change according to the assigned group.
  Arms: verbal explanation group
Other: hand rehabilitation with patient information and exercise forms — hand rehabilitation with patient information and exercise forms
  Arms: patient information and exercise forms group
Other: hand rehabilitation with video recording — hand rehabilitation with video recording
  Arms: video recording group

SUMMARY:
The investigators believe that these information forms, exercise forms and video recordings that provide patient education will contribute to the collaborative approach of the patient and the clinician, the patient's participation in the treatment, the expectation of treatment and results, and their autonomy. The contribution of patient information forms, exercise forms and video recordings, which have become very important in recent years, to different degrees of results will be questioned.

DETAILED DESCRIPTION:
Written and visual information can affect outcome measurements in health care. In addition to verbal information and guidance, written and visual information is also frequently recommended. This information increases patients' clinical knowledge, communication, and satisfaction and reduces potential anxiety.

Forms have been created in various medical fields to inform the patient about medications, applications, and possible risks, and there are many studies on these instruction forms. The effectiveness of patient information forms and exercise forms in physiotherapy and occupational therapy has gained importance in recent years. It is used in areas such as athlete rehabilitation, impingement syndrome, and osteoarthritis.

However, only one study was found, especially in the field of hand rehabilitation.

The aim of planning this study is to examine the contribution of patient information forms, exercise forms, and video recordings to the clinical and functional results of patients who suffered hand and forearm injuries as a result of a work accident.

ELIGIBILITY:
Inclusion Criteria:

* who have a hand or forearm injury as a result of a work-related injury
* who has undergone primary surgery/conservative treatment related to the injury
* who is literate
* who has and can use technological equipment to use visual and audio communication materials (video)

Exclusion Criteria:

* who miss the evaluations
* who wants to leave the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Impact of Event Scale-Revised | The evaluation were completed in the first session when the patient applied to the hand rehabilitation unit, and it was also repeated at 3th months after the surgery or conservative treatment.
  This scale is a 22-item self-report measure that assesses subjective distress caused by traumatic events. Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). The total score ranges from 0 to 88. A higher score indicates more affection for the traumatic event.
State-trait Anxiety Inventory | The evaluation were completed in the first session when the patient applied to the hand rehabilitation unit, and it was also repeated at 3th months after the surgery or conservative treatment.
  This inventory was developed by Spielberger et al. (1970) to measure anxiety from the perspective of states vs. traits. The state measurement assesses how the individual feels "right now" or at this moment. The range of possible scores is from a minimum score of 20 to a maximum score of 80. Scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).

SECONDARY OUTCOMES:
Grip and Pinch Strength | The evaluation were completed in the first session when the patient applied to the hand rehabilitation unit, and it was also repeated at 3th months after the surgery or conservative treatment.
  Grip and Pinch Strength strength is measured in pounds, kilograms by squeezing a dynamometer and a pinchmeter about three times in each hand.
Michigan Hand Outcomes Questionnaire | The evaluation were completed in the first session when the patient applied to the hand rehabilitation unit, and it was also repeated at 3th months after the surgery or conservative treatment.
  This Questionnaire is a tool used to assess patients with hand disorders through the measurement of 6 health domains: overall hand function, activities of daily living, pain, work performance, aesthetics, and patient satisfaction. An overall score can be obtained by summing the scores for all six scales after reversing the pain scale (pain=100-pain score) and then dividing by six. On the pain scale, high scores indicate greater pain, while on the other five scales, high scores denote better hand performance.

CONTACTS AND LOCATIONS:
Overall Officials: ALI KITIS, Professor, Study Director — Pamukkale University Faculty of Physiotherapy and Rehabilitation; AHMET FAHİR DEMIRKAN, Professor, Study Director — Pamukkale University Faculty of Medicine
Locations (1):
- Pamukkale University, Merkez, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abu Abed M, Himmel W, Vormfelde S, Koschack J. Video-assisted patient education to modify behavior: a systematic review. Patient Educ Couns. 2014 Oct;97(1):16-22. doi: 10.1016/j.pec.2014.06.015. Epub 2014 Jul 5. PMID 25043785
- [Background] Barton CJ, Rathleff MS. 'Managing My Patellofemoral Pain': the creation of an education leaflet for patients. BMJ Open Sport Exerc Med. 2016 Mar 31;2(1):e000086. doi: 10.1136/bmjsem-2015-000086. eCollection 2016. PMID 27900163
- [Background] Snyder-Ramos SA, Seintsch H, Bottiger BW, Motsch J, Martin E, Bauer M. Patient satisfaction and information gain after the preanesthetic visit: a comparison of face-to-face interview, brochure, and video. Anesth Analg. 2005 Jun;100(6):1753-1758. doi: 10.1213/01.ANE.0000153010.49776.E5. PMID 15920209